CLINICAL TRIAL: NCT05941416
Title: Evaluation Of Orofacial Myofunctional Disorders Among A Group Of Children With Bronchial Asthma: A Cross-Sectional (Observational) Study
Brief Title: Orofacial Myofunctional Disorder Among Asthmatic Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, yara mamdouh khalifa ahmed, Dentist, Cairo University
Other Study IDs: OMD in Asthmatic
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Orofacial Myofunctional Disorders
Keywords: Orofacial myofunctional disorders; Bronchial Asthma; OMD
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Nordic Orofacial test- screening arabic modified version — Nordic Orofacial Test- screening is an instrument that can be used for the identification of orofacial myofunctional disorders in children aged three years or older, in youths and in adults. It is divided into two sections, interview and examination. The screening can be directed by dental or health care professional personnel.
  Other Names: Child perceptions questionnaire for 8-10-year-old children

SUMMARY:
This study aims to evaluate orofacial myofunctional disorders among a group of children with bronchial asthma.

DETAILED DESCRIPTION:
Scientific Background (Statement of the problem):

Bronchial Asthma is a growing prevalent health problem among pediatric patients. The prevalence of Bronchial Asthma among children and adolescence in Cairo, Egypt was 9.4%. It is a chronic inflammatory disease that affects the lungs characterized by bronchial hyperactivity causing reversible airway obstruction and inflammation, and increased airway receptivity to stimuli. Bronchial Asthma classification, historically, depended on the severity of symptoms, but recently Bronchial Asthma was classified according to levels of control: controlled, partly controlled, or uncontrolled. That recent classification considers not only the disease's severity but also the responsiveness to medications.

As a result of inflammatory response and airway obstruction, difficulty in breathing may cause discomfort to the patients. So oral breathing become an alternative to nasal breathing. This change in the way of breathing can affect craniofacial growth which in sequence affects facial muscles.

The most characteristic features of mouth breathing are a long face, flat nose with narrow nostrils, hypotonic orofacial muscles, and open or semi-open mouth. Early diagnosis of mouth breathing can prevent the development of these features.

The stomatognathic system is a functional complex with a highly adaptable complex of bones, muscles, joints, teeth, lips, tongue, cheeks, glands, arteries, veins, and nerves that act harmoniously. So, any change in this harmony causes imbalance and alteration in the function which is called Orofacial Myofunctional Disorders.

Orofacial Myofunctional Disorders are multifactorial conditions common in many genetic and congenital disorders. As well it can be acquired as a result of mouth breathing, deviate swallowing, TMD, trauma, tongue thrusting, sucking, or chewing habits past the age of 3. Orofacial Myofunctional can be severely disabling as it affects chewing, swallowing, speech, facial expression, appearance and in conclusion affects oral health-related quality of life in children (OHRQoL).

Symptoms of Orofacial Myofunctional Disorders may include facial asymmetry, mouth breathing, tongue thrusting, impaired speech, malocclusion, improper jaw growth, facial pain, drooling, dry mouth and sleeping disorder.

Nordic Orofacial Test- screening (NOT-S) is a comprehensive screening instrument for the assessment of orofacial dysfunction. Nordic Orofacial Test- screening was first reported at the Second Nordic Conference on Orofacial Therapy in Gothenburg in 2002. Nordic Orofacial Test- screening has good reliability and gives a rough discrimination between normal orofacial function and various degrees of orofacial disability.

Oral Health-Related Quality of Life in children (OHRQoL) is determined by social interactions, including speech, emotional communication, facial expression, and appearance. It can be measured by Child Perceptions Questionnaire (CPQ8-10).

This study aims to evaluate orofacial myofunctional disorders among a group of children with Bronchial Asthms

Review of Literature:

Bronchial Asthma is a chronic inflammatory disease that targets millions of children and adolescence on an international scale. In 2006 was reported that the prevalence of Bronchial Asthma was 9.4% among school children and adolescence in Cairo, Egypt. According to the World Health Organization WHO, in 2005, the cost of asthma medication exceeded the cost of AIDS. In 2022, The recent Global Asthma Study (GAN) phase reported that worldwide prevalence of asthma among children reached 11% at age 6-7 years and 9.1 at age 13-14 years.

Bronchial asthma is a lower respiratory tract infection that causes narrowing in bronchial tubes and airway obstruction. It was founded that as a result to airway obstruction, asthmatic patients choose oral breathing as an alternative to nasal breathing.

An association was found between asthma onset and Orofacial Myofunctional Disorders observed in adults. In this study the authors reported that Orofacial Myofunctional Disorders are often observed in asthmatic patients that got affected by the disease before the age of 14. It was also reported that Orofacial Myofunctional Disorders and Malocclusion were found more among asthmatic children and adolescence when compared to healthy children. These children showed inadequate positioning of the jaw and during swallowing of water, tension in the facial muscles was reported Then it was verified that Orofacial Myofunctional Disorders were statistically higher in the asthma group. The highest facial disfunctions had been found were chewing and swallowing food with certain consistency and long mealtime more than 30 minutes. These results affected the Oral Health Quality of Life for the asthmatic patients.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 8-10 years old
* Asthmatic children were selected from the Asthma and Allergy Outpatients Clinic of Abu El-Reesh Japanese Hospital for kids

Exclusion Criteria:

* Children who refused to participate
* Children with Cognitive problems
* Children with neurological diseases
* Children undergoing orthodontic treatment
* Children who underwent speech therapy
* Children who underwent otorhinolaryngology surgery
* Children with a history of oral habits such as thumb sucking, pacifier use, bottle, and nail-biting, over the age of three years

Ages: 8 Years to 10 Years | Sex: All
Age Groups: Child
Study Population: Egyptian children with bronchial asthma aged between 8-10 years old
Sampling Method: Non-Probability Sample
Enrollment: 195 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Orofacial myofunctional disorders | Baseline
  Nordic orofacial test- screening

SECONDARY OUTCOMES:
Oral habits evaluation (Mouth Breathing only) | Baseline
  Massler's water-holding test
Oral Health-Related Quality of Life (OHRQoL) | Baseline
  Children perceptions questionnaire for 8-10-year-old children arabic version (CPQ8-10)

CONTACTS AND LOCATIONS:
Overall Officials: Manal A Elsayed, Professor, Study Director — Cairo University

REFERENCES:
- [Background] Al-Blaihed D, El-Housseiny AA, Farsi NJ, Farsi NM. Validity and reliability of the Arabic version of the child perceptions questionnaire for 8-10-year-old children. Qual Life Res. 2020 Nov;29(11):3131-3141. doi: 10.1007/s11136-020-02545-y. Epub 2020 Jun 10. PMID 32524347
- [Background] Araujo BCL, Lima TRCM, de Gois-Santos VT, Nascimento GKBO, Martins-Filho PR, Simoes SM. Association between nasal patency and orofacial myofunctional changes in patients with asthma and rhinitis. Eur Arch Otorhinolaryngol. 2021 Jul;278(7):2371-2377. doi: 10.1007/s00405-020-06518-2. Epub 2021 Jan 2. PMID 33389007
- [Background] Bakke M, Bergendal B, McAllister A, Sjogreen L, Asten P. Development and evaluation of a comprehensive screening for orofacial dysfunction. Swed Dent J. 2007;31(2):75-84. PMID 17695052
- [Background] Brozek JL, Bousquet J, Agache I, Agarwal A, Bachert C, Bosnic-Anticevich S, Brignardello-Petersen R, Canonica GW, Casale T, Chavannes NH, Correia de Sousa J, Cruz AA, Cuello-Garcia CA, Demoly P, Dykewicz M, Etxeandia-Ikobaltzeta I, Florez ID, Fokkens W, Fonseca J, Hellings PW, Klimek L, Kowalski S, Kuna P, Laisaar KT, Larenas-Linnemann DE, Lodrup Carlsen KC, Manning PJ, Meltzer E, Mullol J, Muraro A, O'Hehir R, Ohta K, Panzner P, Papadopoulos N, Park HS, Passalacqua G, Pawankar R, Price D, Riva JJ, Roldan Y, Ryan D, Sadeghirad B, Samolinski B, Schmid-Grendelmeier P, Sheikh A, Togias A, Valero A, Valiulis A, Valovirta E, Ventresca M, Wallace D, Waserman S, Wickman M, Wiercioch W, Yepes-Nunez JJ, Zhang L, Zhang Y, Zidarn M, Zuberbier T, Schunemann HJ. Allergic Rhinitis and its Impact on Asthma (ARIA) guidelines-2016 revision. J Allergy Clin Immunol. 2017 Oct;140(4):950-958. doi: 10.1016/j.jaci.2017.03.050. Epub 2017 Jun 8. PMID 28602936
- [Background] Castro MS, Toro AA, Sakano E, Ribeiro JD. Evaluation of oral functions of the stomatognathic system according to the levels of asthma severity. J Soc Bras Fonoaudiol. 2012;24(2):119-24. doi: 10.1590/s2179-64912012000200005. English, Portuguese. PMID 22832677
- [Background] D'Onofrio L. Oral dysfunction as a cause of malocclusion. Orthod Craniofac Res. 2019 May;22 Suppl 1(Suppl 1):43-48. doi: 10.1111/ocr.12277. PMID 31074141
- [Background] De Menezes VA, Leal RB, Pessoa RS, Pontes RM. Prevalence and factors related to mouth breathing in school children at the Santo Amaro project-Recife, 2005. Braz J Otorhinolaryngol. 2006 May-Jun;72(3):394-9. doi: 10.1016/s1808-8694(15)30975-7. PMID 17119778
- [Background] Carvalho-Oliveira M, Salles C, Terse R, D'Oliveira A Junior. Association between severe asthma and changes in the stomatognathic system. J Bras Pneumol. 2016 Nov-Dec;42(6):423-428. doi: 10.1590/S1806-37562015000600006. PMID 28117472
- [Background] Garcia-Marcos L, Asher MI, Pearce N, Ellwood E, Bissell K, Chiang CY, El Sony A, Ellwood P, Marks GB, Mortimer K, Martinez-Torres AE, Morales E, Perez-Fernandez V, Robertson S, Rutter CE, Silverwood RJ, Strachan DP; Global Asthma Network Phase I Study Group. The burden of asthma, hay fever and eczema in children in 25 countries: GAN Phase I study. Eur Respir J. 2022 Sep 15;60(3):2102866. doi: 10.1183/13993003.02866-2021. Print 2022 Sep. PMID 35144987
- [Background] Georgy V, Fahim HI, El-Gaafary M, Walters S. Prevalence and socioeconomic associations of asthma and allergic rhinitis in northern [corrected] Africa. Eur Respir J. 2006 Oct;28(4):756-62. doi: 10.1183/09031936.06.00089005. Epub 2006 May 31. PMID 16737986
- [Background] Koshak EA. Classification of asthma according to revised 2006 GINA: evolution from severity to control. Ann Thorac Med. 2007 Apr;2(2):45-6. doi: 10.4103/1817-1737.32228. No abstract available. PMID 19727344
- [Background] de Felicio CM, Melchior Mde O, Ferreira CL, Da Silva MA. Otologic symptoms of temporomandibular disorder and effect of orofacial myofunctional therapy. Cranio. 2008 Apr;26(2):118-25. doi: 10.1179/crn.2008.016. PMID 18468271
- [Background] Milanesi JM, Berwig LC, Marquezan M, Schuch LH, Moraes AB, Silva AMTD, Correa ECR. Variables associated with mouth breathing diagnosis in children based on a multidisciplinary assessment. Codas. 2018 Mar 19;30(4):e20170071. doi: 10.1590/2317-1782/20182017071. PMID 29561967
- [Background] Ukena D, Fishman L, Niebling WB. Bronchial asthma: diagnosis and long-term treatment in adults. Dtsch Arztebl Int. 2008 May;105(21):385-94. doi: 10.3238/arztebl.2008.0385. Epub 2008 May 23. PMID 19626179
- [Background] YILMAZ BC, Alaçam A. Evaluation of orofacial dysfunctions and oral health-related quality of life in children with asthma. Acta Odontologica Turcica. 2023 Jan 1;40(1):22-8.
- [Background] Leme MS, Barbosa TD, Gavião MB. Assessment of orofacial functions in Brazilian children using the Nordic Orofacial Test-Screening (NOT-S). Revista Odonto Ciência. 2012;27:108-14.
- [Background] Cerci Neto A, Kohatsu M, Moreira AC. Programa Respira Londrina. Cerci Neto, A. organizador. Asma em Saúde Pública. São Paulo: Manole. 2007:79-92.